CLINICAL TRIAL: NCT04248530
Title: An Open-Label, Single Arm, Multicenter Feasibility Study to Evaluate the Safety of Catheter-Based Renal Denervation With the DENEX System in Patients With Uncontrolled Hypertension on Standard Medical Therapy
Brief Title: DENEX Renal Denervation in Patients With Uncontrolled Hypertension: Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kalos Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DN_C101
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2020-05

CONDITIONS: Uncontrolled Hypertension
Keywords: Uncontrolled Hypertension; Renal Denervation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal denervation therapy group (Experimental): The subject treated by renal denervation by using DENEX system.
  Interventions: Device: Renal denervation

INTERVENTIONS:
Device: Renal denervation — DENEX catheter is a device to treat resistant hypertension which delivers high-frequency energy through the three electrodes connected to the catheter in order to cauterize sympathetic nerve bundle.

SUMMARY:
The study is the multicenter pilot study to obtain an assessment of the safety of renal denervation in the patients with uncontrolled hypertension on standard medical therapy in Korea.

DETAILED DESCRIPTION:
DENEX system developed by Handok Kalos Medical Inc. is a renal nerve blocking system to efficiently block the sympathetic nerve of the kidney with minimal invasive procedure. It was developed to block the sympathetic nerves distributed in blood vessel wall by delivering high frequency energy to the renal artery for the purpose of treating hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is ≥ 20 years of age at time of consent
2. Individual has office systolic blood pressure (SBP) of ≥ 150 mmHg
3. Individual has daytime 24-hour Ambulatory Blood Pressure Monitoring (ABPM) SBP of ≥ 140 mmHg
4. Individual maintains the following 3 antihypertensive medications: thiazide-type diuretic, calcium-channel blocker, and angiotensin-converting enzyme inhibitor or angiotensin receptor blocker (for at least 6 weeks before the screening visit) that is expected to be maintained without changes for at least 6 months.

Exclusion Criteria:

1. Main renal artery contains renal artery stenosis >50%
2. Individual has confirmed anatomical findings in kidneys or renal arteries through CT scan or angiogram
3. Undergone prior renal angioplasty
4. Main renal arterial vessel for each kidney <4 and >8 mm in diameter, or <20 mm length
5. Individual has an Estimated glomerular filtration rate <45 mL/min/1.73 m2 at screening visit
6. Individual has experienced myocardial infarction, unstable angina pectoris, syncope, or a cerebrovascular accident within 3 months of the screening period, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques
7. Individual has Hemodynamically or echocardiography significant valvular heart disease
8. Individual has secondary hypertension (pheochromocytoma, Cushing syndrome,coarctation of the aorta, renovascular hypertension, primary hyperaldosteronism, or other secondary hypertension)
9. Individual has documented primary pulmonary hypertension
10. Individual has orthostatic hypotension with symptom
11. Individual requires chronic oxygen support for sleep apnea
12. Individual is taking chronic NSAIDs (Non-Steroidal Anti-Inflammatory Drugs). Only, Aspirin is permitted for cardiovascular disease prevention
13. Individual has Type 1 diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Rate of all adverse events | From baseline to 1 month post-procedure
  rate of major adverse events for 1 month after the treatment

SECONDARY OUTCOMES:
Ambulatory SBP change at 3,6,12,24 months | From baseline to 3, 6, 12, 24 months post-procedure
  Change in systolic blood pressure as measured by 24-hour ABPM at 3, 6, 12, 24 months post denervation
Office SBP change at 1, 3, 6, 12, 18, 24 months | From baseline to 1, 3, 6, 12, 18, 24 months post-procedure
  Change in office systolic blood pressure at 1, 3, 6, 12, 18, 24 months post denervation
Percentage of decreased office SBP >10, 15, 20 mmHg | From baseline to 1, 3, 6, 12, 18, 24 months post-procedure
  Percentage of subjects decreased office systolic blood pressure > 10 mmHg, 15 mmHg, 20 mmHg at 1, 3, 6, 12, 18, 24 months post denervation

CONTACTS AND LOCATIONS:
Overall Officials: Yangsu Jang, Principal Investigator — Division of Cardiology, Severance Hospital
Locations (5):
- South Korea (5):
  - Pusan National University Hospital, Pusan
  - Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul St.Mary's Hospital, Seoul
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim CJ, Chang K, Kim BK, Park CG, Jang Y. An Open-label, Single-arm, Multicenter Feasibility Study Evaluating the Safety of Catheter-based Renal Denervation with DENEX in Patients with Uncontrolled Hypertension on Standard Medical Therapy. Korean Circ J. 2021 Jan;51(1):43-55. doi: 10.4070/kcj.2020.0391. PMID 33377328